CLINICAL TRIAL: NCT04373772
Title: The Effect of Abdominal Massage on Bowel Evacuation After Cranial Surgery: A Randomized Controlled Trial
Brief Title: Effect of Abdominal Massage on Bowel Evacuation After Cranial Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gulay ALTUN UGRAS, Associate professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mersin U
Record Dates: First submitted 2020-04-27; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Constipation; Abdominal Massage
Keywords: Cranial surgery; bowel evacuation; constipation; abdominal massage; nursing
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: prospective, parallel, two arm (1:1), randomized controlled clinical trial
Who Masked: Participant
Masking Description: In this study, due to the nature of the intervention, only the patient was blinded. The researchers involved in the running of the study were not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- abdominal massage group (Experimental): the abdominal massage group received a total of 30 minutes of massage, 15 minutes every morning and evening, until the first defecation.
  Interventions: Other: abdominal massage
- control group (No Intervention): Routine care for the control group

INTERVENTIONS:
Other: abdominal massage — the patients in the AM group were given a total of 30 minutes of AM by the nurses (HD, OM) everyday for 15 minutes in the morning and evening.In this study AM, which included effleurage, strokes, petrissage and vibration techniques, was applied to the patients for 15 minutes in each session at 9:00 am and 9:00 pm.
  Arms: abdominal massage group

SUMMARY:
Many factors in patients undergoing cranial surgery (CS) may affect the bowel evacuation of patients, resulting in constipation, which could lead to the use of the valsalva maneuver. The aim of this study was to determine the effect of abdominal massage (AM) on bowel evacuation of patients treated in intensive care units (ICU) after CS.

DETAILED DESCRIPTION:
The sample of this prospective parallel two-arm randomized controlled trial included 80 patients who underwent CS. The patients were randomly assigned (1:1) to the AM and control groups. The constipation risk of all the patients following CS was assessed with Constipation Risk Assessment Scale (CRAS). Those patients in the AM group received a total of 30 minutes of massage, 15 minutes every morning and evening, until the first defecation. The bowel sounds of all the patients in the AM and control groups were assessed on a daily basis. The days when bowel sounds were heard and the first defecation took place were recorded in a Bowel Evacuation Form.

ELIGIBILITY:
Inclusion Criteria: Patients who

* volunteered to participate in the study,
* were 18 years old or older and underwent CS,
* stayed in the ICU for ≥ 3 days,

Exclusion Criteria: Patients who

* have percutaneous endoscopic gastrostomy,
* abdominal hernia,
* irritable bowel syndrome
* bowel cancer,
* history of abdominal surgery,
* pregnancy,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — ≥18 years old
Enrollment: 80 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Primery outcome: bowel sounds | up to 10 days
  time return of bowel sounds
Primery outcome: first defecation | up to 10 days
  time of the first defecation

SECONDARY OUTCOMES:
constipation risk | up to 24 hours
  constipation risk in intensive care unit